CLINICAL TRIAL: NCT05615636
Title: A Phase II Trial of Mosunetuzumab, Polatuzumab, Tafasitamab, and Lenalidomide in Patients With Relapsed B-cell NHL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0459; NCI-2022-09576 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hodgkin Lymphoma; B-Cell Lymphoma; Relapsed B-cell NHL
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, B-Cell | interventions — polatuzumab vedotin; tafasitamab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety Run In (Experimental): During the safety run-in, the study team will first test a recommended dose of mosunetuzumab, polatuzumab vedotin, tafasitamab, and lenalidomide.
  Interventions: Drug: Mosunetuzumab; Drug: Polatuzumab vedotin; Drug: Tafasitamab; Drug: Lenalidomide
- Dose Expansion Cohort (Experimental): Participants will receive mosunetuzumab, polatuzumab vedotin, tafasitamab, and lenalidomide at the dose level that was found tolerated in the safety run-in.
  Interventions: Drug: Mosunetuzumab; Drug: Polatuzumab vedotin; Drug: Tafasitamab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Mosunetuzumab — Given by IV (vein)
  Other Names: RO7030816
Drug: Polatuzumab vedotin — Given by IV (vein)
Drug: Tafasitamab — Given by IV (vein)
Drug: Lenalidomide — Given by PO
  Other Names: CC-5013; Revlimid

SUMMARY:
To learn if giving mosunetuzumab in combination with polatuzumab vedotin, tafasitamab, and lenalidomide can help to control relapsed/refractory FL and DLBCL.

DETAILED DESCRIPTION:
Primary Objectives:

To determine the safety of mosunetuzumab, polatuzumab vedotin, tafasitamab, and lenalidomide in relapsed/refractory NHL.

To determine the best overall response rate (ORR) of the combination of mosunetuzumab, with polatuzumab vedotin, tafasitamab, and lenalidomide in patients with relapsed/refractory diffuse large B-cell lymphoma.

Secondary Objectives:

To determine the complete response rate, duration of response, progression free survival, and overall survival in patients with DLBCL following treatment with of mosunetuzumab, polatuzumab vedotin, tafasitamab, and lenalidomide.

To evaluate changes in immune effector cells and the tumor microenvironment following treatment with of mosunetuzumab, polatuzumab vedotin, tafasitamab, and lenalidomide.

ELIGIBILITY:
Inclusion criteria:

Patients in safety run in must meet the following criteria for study entry:

* A diagnosis of relapsed CD20+ Follicular Lymphoma grade 1-3a
* A diagnosis of relapsed CD20+ diffuse large B-cell lymphoma

Patients in dose expansion must meet the following criteria for study entry:

• A diagnosis of relapsed CD20+ diffuse large B-cell lymphoma

Patients in each component (safety run in and dose expansion) must meet the following criteria for study entry:

1. Evidence of progression or lack of response following at least 1 prior treatment
2. Able and willing to provide written informed consent and to comply with the study protocol
3. Age ≥ 18 years as these drugs have not yet established safety and efficacy in pediatric patients
4. At least 1 node greater than 1.5cm in short axis diameter
5. Adequate hematologic function (unless abnormalities are related to NHL), defined as follows:

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count ≥ 1.0 x 109/L
   * Platelet count ≥ 75 x 109/L
6. Serum bilirubin <1.5x ULN except in patients with Gilbert's syndrome as defined by > 80% unconjugated bilirubin who must have a serum bilirubin of <4x ULN; AST (SGOT) and ALT (SGPT) ≤ 3x ULN or < 5x ULN if hepatic metastases are present
7. Renal function assessed by calculated creatinine clearance:

   • Calculated creatinine clearance ≥ 30ml/min by Cockcroft-Gault formula. See section below, "Dosing Regimen", regarding lenalidomide dose adjustment for calculated creatinine clearance ≥ 30ml/min and < 60ml/min.
8. Patients must be willing to receive transfusions of blood products.
9. For men who are not surgically sterile, agreement to use a barrier method of contraception for ≥ 3 months after the last treatment dose. In addition, male patients must agree to request that their partners use an additional method of contraception, such as oral contraceptives, intrauterine device, barrier method of contraception, or spermicidal jelly. With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for 60 days after the final dose of mosunetuzumab, 6 months after the final dose of polatuzumab vedotin, and 60 days after the final dose of tocilizumab, as applicable, to avoid exposing the embryo. Men must refrain from donating sperm during this same period.
10. For women of reproductive potential who are not surgically sterile, agreement to use two adequate methods of contraception, such as oral contraceptives, intrauterine device, or barrier method of contraception in conjunction with spermicidal jelly for≥ 12 months after the last therapeutic drug dose
11. Females of childbearing potential (FCBP, defined as a female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2)has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months). must have a negative serum pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a female of childbearing potential even if they have had a successful vasectomy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women must refrain from donating eggs during this same period.
12. All study participants must be registered into the mandatory Revlimid REMS® program and be willing and able to comply with the requirements of Revlimid REMS® program.
13. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).

Exclusion Criteria:

1. Known hypersensitivity to any study drug
2. Prior treatment with polatuzumab vedotin
3. Prior treatment with mosunetuzumab or other CD20-directed bispecific antibodies
4. Prior treatment with tafasitamab and/or lenalidomide
5. Autologous SCT within 100 days prior to first study treatment administration
6. Prior treatment with CAR-T therapy within 30 days before first study treatment administration
7. Current eligibility for autologous SCT in patients with R/R DLBCL
8. Prior allogeneic SCT
9. Prior solid organ transplantation
10. History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
11. Regular treatment with corticosteroids during the 2 weeks prior to the start of Cycle 1, unless administered for indications other than NHL at a dose equivalent to < 20 mg/day prednisone. Treatment with systemic immunosuppressive medications, including, but not limited to, prednisone (20 mg), azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents within 2 weeks prior to Day 1 of Cycle 1. The use of inhaled corticosteroids is permitted The use of mineralocorticoids for management of orthostatic hypotension is permitted. Single dose of dexamethasone for nausea or B symptoms is permitted
12. Prior systemic treatment with chemotherapy, immunotherapy, targeted and biologic therapy 4 weeks prior to C1D1.
13. Prior treatment with radiotherapy within 2 weeks prior to C1D1. If patients have received radiotherapy within 4 weeks prior to the initiation of study treatment, patients must have at least one measurable lesion outside of the radiation field. Patients who have only one measurable lesion that was previously irradiated but subsequently progressed are eligible.
14. History of prior malignancy within the last 2 years, except for curatively treated basal or squamous cell carcinoma of the skin and low- grade in situ carcinoma of the cervix
15. Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results including but not limited to uncontrolled hypertension, uncontrolled congestive heart failure within past 6 months prior to screening (Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification), uncontrolled or symptomatic arrhythmias with corrected QT interval (QTc) > 480 msec at screening, uncontrolled diabetes mellitus, active/symptomatic coronary artery disease, COPD, LVEF less than 40%, renal failure, uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura active infection, history of invasive fungal infection, moderate to severe hepatic disease (Child Pugh Class B or C), active hemorrhage, laboratory abnormality, or psychiatric illness that, in the investigators opinion places the patient at unacceptable risk and would prevent the subject from signing the informed consent form. Patients with history of cardiac arrhythmias should have cardiac evaluation and clearance.
16. Known or suspected history of hemophagocytic lymphohistiocytosis
17. History of autoimmune disease, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study. Patients with a history of disease-related immune thrombocytopenic purpura, autoimmune hemolytic anemia, or other stable autoimmune diseases may be eligible after review and approval by the Medical Monitor.
18. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics, except if for tumor fever) within 2 weeks prior to the start of cycle 1
19. Patients with suspected active or latent tuberculosis (latent tuberculosis needs to be confirmed by positive Interferon-gamma release assay)
20. Known or suspected chronic active Epstein-Barr virus (EBV) infection
21. Known HIV infection. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antigen (HBsAg) negative will need to have a negative DNA polymerase chain reaction (PCR) and must be willing to undergo DNA PCR testing during the study to be eligible. Those who are HBsAg positive or hepatitis B DNA PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative DNA PCR result to be eligible. Those who are hepatitis C DNA PCR positive will be excluded.
22. Vaccination with live vaccines within 28 days prior to start of treatment
23. No peripheral neuropathy ≥ grade 2 or = grade 2 with pain
24. Pregnant or lactating females.
25. All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
26. Women of childbearing potential must have a negative serum (-human chorionic gonadotropin [-hCG]) at screening and must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
27. All patients with known central nervous system involvement with lymphoma.
28. Contraindication to any of the required concomitant drugs or supportive treatments or intolerance to hydration due to preexisting pulmonary or cardiac impairment including pleural effusion requiring thoracentesis or ascites requiring paracentesis not due to lymphoma.
29. Patients with active pulmonary embolism or deep vein thrombosis (diagnosed within 30 days of study enrollment).
30. Major surgery within 4 weeks of study entry, or wound that is not healed from prior surgery or trauma.
31. History of stroke or intracranial hemorrhage within 6 months prior to study entry.
32. Active bleeding or history of bleeding diathesis (eg, hemophilia or von Willebrand disease).
33. Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura).
34. Prothrombin time (PT)/INR or aPTT (in the absence of lupus anticoagulant) >2x ULN.
35. Concurrent participation in another therapeutic clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2027-08-19 (Estimated); Study Completion 2027-08-19 (Estimated)

PRIMARY OUTCOMES:
The best overall response rate (ORR). | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Westin, MD, MS, FACP, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-12-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT05615636/ICF_000.pdf